CLINICAL TRIAL: NCT02342548
Title: An Open Label Extension Study To Investigate The Long Term Safety, Tolerability And Efficacy Of Pf-02545920 In Subjects With Huntington's Disease Who Previously Completed Study A8241021
Brief Title: Open Label Extension Study To Investigate Long Term Safety, Tolerability And Efficacy Of Pf-02545920 In Subjects With Huntington's Disease Who Completed Study A8241021
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated on 15DEC2016 due to study A8241021 showing no significant difference on primary endpoint between PF-02545920 & placebo. No safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8241022; 2014-004900-31 (EudraCT Number); OPEN LABEL TO A8241021 (Other: Alias Study Number)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Huntington's Disease
Keywords: Huntington; chorea; total motor score; CAG repeat: total functional capacity; motor cognitive and behavioral symptoms
MeSH Terms: conditions — Huntington Disease; Chorea; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 mg BID PF-02545920 non-titrated (Experimental): Subjects who received 20 mg BID in completed study A8241021 will continue to receive 20 mg BID PF-02545920
  Interventions: Drug: 20 mg BID of PF-02545920
- 20mg BID PF-02545920 titrated (Experimental): Subjects who received either Placebo or 5mg BID of PF-02545920 in completed study A8241021 will be titrated up to 20 mg with 5mg increment per week, over 4 weeks (5mg increment/wk)
  Interventions: Drug: 20 mg BID of PF-02545920

INTERVENTIONS:
Drug: 20 mg BID of PF-02545920 — All subject who completed A8241021 will receive 20 mg BID (with or without titration)

SUMMARY:
This study is a 12 month open label extension study of PF-02545920 20 mg dosed BID following study A8241021 in subjects with HD. Primary endpoints will be to assess long-term safety and tolerability of 20 mg BID of PF-02545920. Secondary endpoints will be the change from baseline in the Total Motor Score (TMS)assessment, and/ior the Total maximum Chorea (TMC) assessment of the Unified Huntington Disease Rating Scale (UHDRS) after 6 and 12 months of treatment, and Clinical Global Impression-Improvement score after 6 and 12 months of treatment. Subjects, who were assigned to the 20 mg PF-02545920 dose group in the preceding A8241021 study, will receive 20 mg PF-02545920 without any titration. All other subjects will be titrated to the 20 mg BID dose as follows: 5 mg BID for 7 days, 10 mg BID for 7 days, 15 mg BID for 7 days, then 20 mg BID for the remainder of the treatment phase. Up to 260 subjects may take part in this open label extension

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed study A8241021
* Diagnosis of HD, including ≥36 CAG repeats.

Exclusion Criteria:

* Significant neurological disorder other than Huntington's disease.
* WBC ≤ 3500/mm3 AND/OR ANC ≤ 2000/mm3 and history of neutropenia or myeolo-proliferative disorders.
* Any drug related SAE experienced during study A8241021 which were not approved as acceptable for enrollment in A8241022.

Ages: 30 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (17):
  - The Kirkland Clinic of UAB Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Ronald Reagan UCLA Medical Center Drug Information Center, Los Angeles, California
  - UCLA Neurology Clinic, Los Angeles, California
  - UCLA Radiology, Los Angeles, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - University of Florida Center for Movement Disorders & Neurorestoration, Gainesville, Florida
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - The Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - The Wright Center of Innovation- The Ohio State University, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
- Canada (4):
  - The Centre For Huntington Disease, The University of British Columbia, Vancouver, British Columbia
  - Center For Movement Disorders, Toronto, Ontario
  - CHUM-Notre-Dame Hospital, Montreal, Quebec
  - CHUM-Notre-Dame, Pharmacie, Montreal, Quebec
- Germany (11):
  - Uniklinik RWTH Aachen, Aachen
  - Charité - Universitätsmedizin Berlin, Berlin
  - St. Josef Hospital, Bochum
  - Friedrich-Alexander-Universität, Erlangen
  - Universität zu Lübeck, Lübeck
  - Philipps Universitat Marburg, Marburg
  - Technische Universität München, München
  - George-Huntington-Institut, Münster
  - Kbo-Isar-Amper-Klinikum gGmbH, Taufkirchen
  - Universitätsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Poland (4):
  - Copernicus Podmiot Leczniczy sp.zo.o, Gdansk
  - Krakowska Akademia Neurologii Sp. zo.o, Krakow
  - Solumed Centrum Medyczne, Poznan
  - Instytut Psychiatrii i Neurologii, I Klinika Neurologiczna, Warsaw
- United Kingdom (14):
  - Central Manchester University Hospitals NHS Foundation Trust, Oxford Road, Manchester
  - St Nicholas Hospital, Gosforth, Newcastle UPON TYNE
  - Bimingham & Solihull Mental Health NHS Foundation Trust Department of Neuropsychiatry, Birmingham, WEST Midlands
  - NHS Grampian, Aberdeen Royal Infirmary, Clinical Genetics Centre, Aberdeen
  - Institute of Psychological Medicine and Clinical Neurosciences, Cardiff
  - NHS Greater Glasgow and Clyde, Glasgow
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - University College London Hospitals Huntington's Diesease, London
  - University College London Hospitals NHS Foundation Trust, London
  - The National Institute for Health Research / Wellcome Trust Clinical Research Facility, Manchester
  - Newcastle Magnetic Resonance Centre, Newcastle upon Tyne
  - Oxford University Hospitals NHS Trust, Oxford
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Wessex Neurological Centre, Southampton

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241022&StudyName=An%20Open%20Label%20Extension%20Study%20To%20Investigate%20The%20Long%20Term%20Safety%2C%20Tolerability%20And%20Efficacy%20Of%20Pf-02545920%20In%20Subjects%20With%20Huntington%E2%80%99s%20Disease%20Who%20Previously%20Completed%20Study%20A8241021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label extension study conducted in participants who had completed study A8241021 (NCT02197130). Treatment assignment was double-blinded from Day 1 to Day 21, and became open-label from Day 22, since all participants began receiving the same dose level from Day 22.
Groups:
- 20 mg PF-02545920: Participants who received PF-02545920 20 mg twice daily (BID) in Study A8241021 continued to receive PF-02545920 20 mg BID for 12 months in this study. Four 5-mg tablets were administered orally each time.
- 5 mg PF-02545920 Titration up to 20 mg: Participants who received PF-02545920 5 mg twice daily (BID) in Study A8241021 were administered PF-02545920 orally according to a double-blind titration schedule in this study: 5 mg BID for 7 days (one 5-mg tablet and 3 placebo tablets); 10 mg BID for 7 days (two 5-mg tablets and 2 placebo tablets); 15 mg BID for 7 days (three 5-mg tablets and 1 placebo tablet); 20 mg BID to Month 12 (four 5-mg tablets).
- Placebo and Titration up to 20 mg PF-02545920: Participants who received placebo twice daily (BID) in Study A8241021 were administered PF-02545920 orally according to a double-blind titration schedule in this study: 5 mg BID for 7 days (one 5-mg tablet and 3 placebo tablets); 10 mg BID for 7 days (two 5-mg tablets and 2 placebo tablets); 15 mg BID for 7 days (three 5-mg tablets and 1 placebo tablet); 20 mg BID to Month 12 (four 5-mg tablets).
Period: Overall Study
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Started | 51 | 71 | 66
Completed | 17 | 9 | 23
Not Completed | 34 | 62 | 43
Not completed — Adverse Event | 12 | 17 | 13
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Study terminated by sponsor | 20 | 39 | 25
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920 | Total
Number analyzed (Participants) | 51 | 71 | 66 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.4) | 48.4 (8.6) | 51.3 (9.4) | 49.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 43 | 101
  Male | 26 | 38 | 23 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White | 50 | 68 | 66 | 184
  Other | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of its causal relationship with study treatment. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; was life-threatening (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study treatment and up to 28 calendar days after the last administration of study treatment that were absent before treatment or that worsened after treatment. AEs included both serious and non-serious AEs.
Time Frame: 1 year
Population: Safety analysis population included all participants who entered the extension study with at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants
  AEs | 39 | 63 | 62
  SAEs | 7 | 9 | 5

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: The laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, absolute total neutrophils, eosinophils, monocytes, basophils, and lymphocytes), chemistry (blood urea nitrogen/urea, creatinine, glucose, glycosylated hemoglobin [diabetics only], calcium, phosphorus, magnesium, creatine kinase, sodium, potassium, chloride, total carbon dioxide, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein), urinalysis (color, appearance, specific gravity, pH, qualitative glucose, qualitative protein, qualitative blood, ketones, nitrites, leukocyte esterase, and microscopy), and other tests (follicle stimulating hormone, urine drug screen, urine pregnancy [human chorionic gonadotropin, hCG], serum beta hCG). Abnormality was determined by the investigator.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants | 19 | 27 | 28

3. Primary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Summarization Criteria
Description: Number of participants with vital signs data meeting the following criteria is presented: (1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); (2) standing SBP <90 mmHg; (3) supine diastolic blood pressure (DBP) <50 mmHg; (4) standing DBP <50 mmHg; (5) supine pulse rate <40 beats per minute (bpm); (6) supine pulse rate >120 bpm; (7) standing pulse rate <40 bpm; (8) standing pulse rate >140 bpm; (9) maximum increase from baseline in supine SBP >= 30 mmHg; (10) maximum increase from baseline in standing SBP >= 30 mmHg; (11) maximum increase from baseline in supine DBP >= 20 mmHg; (12) maximum increase from baseline in standing DBP >= 20 mmHg; (13) maximum decrease from baseline in supine SBP >=30 mmHg; (14) maximum decrease from baseline in standing SBP >=30 mmHg; (15) maximum decrease from baseline in supine DBP >=20 mmHg; (16) maximum decrease from baseline in standing DBP >=20 mmHg.
Time Frame: 1 year
Population: The analysis population included all participants who entered the extension study with at least 1 dose of study medication, and with available data for at least 1 category.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants
  Supine SBP <90 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine SBP <90 mmHg | 0 | 0 | 0
  Standing SBP <90 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Standing SBP <90 mmHg | 0 | 1 | 0
  Supine DBP <50 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine DBP <50 mmHg | 0 | 1 | 0
  Standing DBP <50 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Standing DBP <50 mmHg | 0 | 1 | 0
  Supine pulse rate <40 bpm: number analyzed (Participants) | 49 | 69 | 65
  Supine pulse rate <40 bpm | 0 | 0 | 0
  Supine pulse rate >120 bpm: number analyzed (Participants) | 49 | 69 | 65
  Supine pulse rate >120 bpm | 0 | 0 | 0
  Standing pulse rate <40 bpm: number analyzed (Participants) | 49 | 69 | 65
  Standing pulse rate <40 bpm | 0 | 0 | 0
  Standing pulse rate >140 bpm: number analyzed (Participants) | 49 | 69 | 65
  Standing pulse rate >140 bpm | 0 | 0 | 0
  Supine SBP increase from baseline >=30 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine SBP increase from baseline >=30 mmHg | 3 | 1 | 6
  Standing SBP increase from baseline >=30 mmHg: number analyzed (Participants) | 48 | 69 | 64
  Standing SBP increase from baseline >=30 mmHg | 1 | 6 | 4
  Supine DBP increase from baseline >=20 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine DBP increase from baseline >=20 mmHg | 4 | 2 | 6
  Standing DBP increase from baseline >=20 mmHg: number analyzed (Participants) | 48 | 69 | 64
  Standing DBP increase from baseline >=20 mmHg | 3 | 8 | 2
  Supine SBP decrease from baseline >=30 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine SBP decrease from baseline >=30 mmHg | 2 | 1 | 4
  Standing SBP decrease from baseline >=30 mmHg: number analyzed (Participants) | 48 | 69 | 64
  Standing SBP decrease from baseline >=30 mmHg | 0 | 1 | 2
  Supine DBP decrease from baseline >=20 mmHg: number analyzed (Participants) | 49 | 69 | 65
  Supine DBP decrease from baseline >=20 mmHg | 0 | 2 | 7
  Standing DBP decrease from baseline >=20 mmHg: number analyzed (Participants) | 48 | 69 | 64
  Standing DBP decrease from baseline >=20 mmHg | 1 | 4 | 6

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Categorical Summarization Criteria
Description: Maximum absolute values and increases from baseline were summarized for PR interval (interval between the start of the ECG P wave and the start of the QRS complex corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization), QRS complex (time from Q wave to the end of the S wave corresponding to ventricular depolarization), and QTcF interval (time from ECG Q wave to the end of T wave corresponding to electrical systole, corrected for heart rate using Fridericia's formula). Number of participants with ECG data meeting the following criteria is presented: (1) PR interval >=300 msec; (2) QRS complex >=140 msec; (3) QTcF interval: 450 to <480 msec; (4) QTcF interval: 480 to <500 msec; (5) QTcF interval >=500 msec; (6) PR interval increase from baseline >=25/50 percent; (7) QRS complex increase from baseline >=50 percent; (8) QTcF interval increase from baseline: 30 to <60 msec; (9) QTcF interval increase from baseline >=60 msec.
Time Frame: 1 year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants
  PR interval >=300 msec: number analyzed (Participants) | 50 | 69 | 66
  PR interval >=300 msec | 0 | 0 | 0
  QRS complex >=140 msec: number analyzed (Participants) | 50 | 69 | 66
  QRS complex >=140 msec | 0 | 0 | 0
  QTcF interval: 450 to <480 msec: number analyzed (Participants) | 50 | 69 | 66
  QTcF interval: 450 to <480 msec | 2 | 2 | 2
  QTcF interval: 480 to <500 msec: number analyzed (Participants) | 50 | 69 | 66
  QTcF interval: 480 to <500 msec | 0 | 0 | 1
  QTcF interval >=500 msec: number analyzed (Participants) | 50 | 69 | 66
  QTcF interval >=500 msec | 0 | 0 | 0
  PR interval increase from baseline >=25/50 percent: number analyzed (Participants) | 50 | 66 | 66
  PR interval increase from baseline >=25/50 percent | 0 | 0 | 0
  QRS complex increase from baseline >=50 percent: number analyzed (Participants) | 50 | 66 | 66
  QRS complex increase from baseline >=50 percent | 0 | 0 | 0
  QTcF increase from baseline: 30 to <60 msec: number analyzed (Participants) | 50 | 66 | 66
  QTcF increase from baseline: 30 to <60 msec | 3 | 5 | 4
  QTcF increase from baseline >=60 msec: number analyzed (Participants) | 50 | 66 | 66
  QTcF increase from baseline >=60 msec | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal White Blood Cell Count and Absolute Neutrophil Count (Without Regard to Baseline Abnormality)
Description: Number of participants with white blood cell (WBC) count and absolute neutrophil count (ANC) meeting the following criteria is presented: (1) WBC count <0.6 *the lower limit of normal (LLN); (2) WBC count >1.5 times the upper limit of normal (ULN); (3) ANC <0.8*LLN; and (4) ANC >1.2*ULN.
Time Frame: 1 year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 65
Participants
  WBC < 0.6*LLN | 0 | 0 | 0
  WBC > 1.5*ULN | 1 | 0 | 1
  ANC < 0.8*LLN | 1 | 0 | 0
  ANC > 1.2*ULN | 3 | 4 | 7

6. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Normal Baseline)
Description: as for outcome 2
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants | 13 | 22 | 23

7. Primary Outcome: Number of Participants With Adverse Events Related to Extrapyramidal Symptoms by Severity
Description: Adverse events related to extrapyramidal symptoms included dystonia, akathisia, tardive dyskinesia). Severity was assessed by the investigator. Mild means the AE didn't interfere with the participant's usual function. Moderate means the AE interfered to some extent the participant's usual function. Severe means the AE interfered significantly with the participant's usual function.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants
  Mild dystonia | 0 | 1 | 0
  Moderate dystonia | 0 | 1 | 1
  Severe dystonia | 0 | 0 | 0
  Mild akathisia | 1 | 1 | 0
  Moderate akathisia | 0 | 1 | 3
  Severe akathisia | 0 | 0 | 1
  Mild dyskinesia | 0 | 2 | 4
  Moderate dyskinesia | 1 | 1 | 2
  Severe dyskinesia | 0 | 0 | 0

8. Primary Outcome: Number of Participants in Each Columbia Classification Algorithm of Suicide Assessment (C-CASA) Category
Description: Columbia Suicide Severity Rating Scale (C-SSRS) was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior, and was used in this study. C-SSRS responses were mapped onto the Columbia Classification Algorithm of Suicide Assessment (C-CASA). Number of participants with any of the following behaviors occurring since last visit was summarized: completed suicide; suicide attempt; preparatory acts towards suicide; suicidal ideation; self-injurious behavior (no suicidal intent).
Time Frame: Baseline (Day 1), Weeks 2 and 4, Months 3, 6, 9 and 12, follow-up visit (7-14 days after the last dose of Month 12)
Population: The analysis population included all participants who entered the extension study with at least 1 dose of study medication, and with available data for at least 1 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 51 | 71 | 66
Participants
  Day 1: completed suicide | 0 | 0 | 0
  Day 1: suicide attempt | 0 | 0 | 0
  Day 1: preparatory acts towards suicide | 0 | 0 | 0
  Day 1: suicidal ideation | 0 | 1 | 1
  Day 1: self-injurious behavior | 0 | 0 | 0
  Week 2: completed suicide: number analyzed (Participants) | 51 | 69 | 64
  Week 2: completed suicide | 0 | 0 | 0
  Week 2: suicide attempt: number analyzed (Participants) | 51 | 69 | 64
  Week 2: suicide attempt | 0 | 0 | 0
  Week 2: preparatory acts towards suicide: number analyzed (Participants) | 51 | 69 | 64
  Week 2: preparatory acts towards suicide | 0 | 0 | 0
  Week 2: suicidal ideation: number analyzed (Participants) | 51 | 69 | 64
  Week 2: suicidal ideation | 0 | 0 | 1
  Week 2: self-injurious behavior: number analyzed (Participants) | 51 | 69 | 64
  Week 2: self-injurious behavior | 0 | 0 | 0
  Week 4: completed suicide: number analyzed (Participants) | 50 | 66 | 63
  Week 4: completed suicide | 0 | 0 | 0
  Week 4: suicide attempt: number analyzed (Participants) | 50 | 66 | 63
  Week 4: suicide attempt | 0 | 0 | 0
  Week 4: preparatory acts towards suicide: number analyzed (Participants) | 50 | 66 | 63
  Week 4: preparatory acts towards suicide | 0 | 0 | 0
  Week 4: suicidal ideation: number analyzed (Participants) | 50 | 66 | 63
  Week 4: suicidal ideation | 0 | 1 | 1
  Week 4: self-injurious behavior: number analyzed (Participants) | 50 | 66 | 63
  Week 4: self-injurious behavior | 0 | 0 | 0
  Month 3: completed suicide: number analyzed (Participants) | 42 | 61 | 57
  Month 3: completed suicide | 0 | 0 | 0
  Month 3: suicide attempt: number analyzed (Participants) | 42 | 61 | 57
  Month 3: suicide attempt | 0 | 0 | 0
  Month 3: preparatory acts towards suicide: number analyzed (Participants) | 42 | 61 | 57
  Month 3: preparatory acts towards suicide | 0 | 0 | 0
  Month 3: suicidal ideation: number analyzed (Participants) | 42 | 61 | 57
  Month 3: suicidal ideation | 1 | 0 | 1
  Month 3: self-injurious behavior: number analyzed (Participants) | 42 | 61 | 57
  Month 3: self-injurious behavior | 0 | 0 | 0
  Month 6: completed suicide: number analyzed (Participants) | 35 | 37 | 42
  Month 6: completed suicide | 0 | 0 | 0
  Month 6: suicide attempt: number analyzed (Participants) | 35 | 37 | 42
  Month 6: suicide attempt | 0 | 0 | 0
  Month 6: preparatory acts towards suicide: number analyzed (Participants) | 35 | 37 | 42
  Month 6: preparatory acts towards suicide | 0 | 0 | 0
  Month 6: suicidal ideation: number analyzed (Participants) | 35 | 37 | 42
  Month 6: suicidal ideation | 1 | 0 | 1
  Month 6: self-injurious behavior: number analyzed (Participants) | 35 | 37 | 42
  Month 6: self-injurious behavior | 0 | 0 | 0
  Month 9: completed suicide: number analyzed (Participants) | 26 | 20 | 29
  Month 9: completed suicide | 0 | 0 | 0
  Month 9: suicide attempt: number analyzed (Participants) | 26 | 20 | 29
  Month 9: suicide attempt | 0 | 0 | 0
  Month 9: preparatory acts towards suicide: number analyzed (Participants) | 26 | 20 | 29
  Month 9: preparatory acts towards suicide | 0 | 0 | 0
  Month 9: suicidal ideation: number analyzed (Participants) | 26 | 20 | 29
  Month 9: suicidal ideation | 0 | 1 | 0
  Month 9: self-injurious behavior: number analyzed (Participants) | 26 | 20 | 29
  Month 9: self-injurious behavior | 0 | 0 | 0
  Month 12: completed suicide: number analyzed (Participants) | 48 | 69 | 65
  Month 12: completed suicide | 0 | 0 | 0
  Month 12: suicide attempt: number analyzed (Participants) | 48 | 69 | 65
  Month 12: suicide attempt | 1 | 0 | 0
  Month 12: preparatory acts towards suicide: number analyzed (Participants) | 48 | 69 | 65
  Month 12: preparatory acts towards suicide | 1 | 0 | 0
  Month 12: suicidal ideation: number analyzed (Participants) | 48 | 69 | 65
  Month 12: suicidal ideation | 3 | 0 | 3
  Month 12: self-injurious behavior: number analyzed (Participants) | 48 | 69 | 65
  Month 12: self-injurious behavior | 1 | 0 | 0
  Follow up: completed suicide: number analyzed (Participants) | 23 | 13 | 26
  Follow up: completed suicide | 0 | 0 | 0
  Follow up: suicide attempt: number analyzed (Participants) | 23 | 13 | 26
  Follow up: suicide attempt | 0 | 0 | 0
  Follow up: preparatory acts towards suicide: number analyzed (Participants) | 23 | 13 | 26
  Follow up: preparatory acts towards suicide | 0 | 0 | 0
  Follow up: suicidal ideation: number analyzed (Participants) | 23 | 13 | 26
  Follow up: suicidal ideation | 1 | 0 | 0
  Follow up: self-injurious behavior: number analyzed (Participants) | 23 | 13 | 26
  Follow up: self-injurious behavior | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score
Description: The UHDRS is a clinical rating scale developed to provide a uniform assessment of the clinical features and course of Huntington's disease (HD). The components of the full UHDRS assess motor function, cognition, behavior and functional abilities. Total Motor Score (TMS) assesses motor features of HD with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural ability. The total motor impairment scores was the sum of all the individual 31 motor sub-items (each rated from 0 to 4), with higher scores indicating more severe motor impairment than lower scores. The range of TMS is 0-124.
Time Frame: Baseline (Day 1), Month 6, and Month 12
Population: Full analysis set (FAS) included all participants who had an open-label extension study baseline efficacy evaluation and completed at least Week 2 visit with a valid UHDRS TMS score, and took >=1 dose of open-label study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 50 | 70 | 62
units on a scale
  Month 6: number analyzed (Participants) | 33 | 39 | 40
  Month 6 | 2.4 (7.21) | 3.5 (7.61) | 0.7 (7.43)
  Month 12: number analyzed (Participants) | 15 | 9 | 22
  Month 12 | 4.9 (10.17) | 3.3 (6.71) | 0.6 (8.24)

10. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Maximum Chorea (TMC) Score
Description: The UHDRS is a clinical rating scale developed to provide a uniform assessment of the clinical features and course of Huntington's disease (HD). The components of the full UHDRS assess motor function, cognition, behavior and functional abilities. Total Maximum Chorea (TMC) is a subset of the TMS assessment, and composed of the scoring of 7 chorea assessments (face, orobuccolingual, trunk, right and left upper extremities, right and left lower extremities). Each assessment is rated from 0 to 4 (absent to prolonged). TMC is obtained by adding up each of the separate scores, leading to max score of 28. The minimum score is 0. The higher the score, the worse the symptoms.
Time Frame: Baseline (Day 1), Month 6, and Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 50 | 70 | 62
Units on a scale
  Month 6: number analyzed (Participants) | 33 | 39 | 40
  Month 6 | 0.1 (3.12) | 1.3 (3.97) | 1.4 (4.14)
  Month 12: number analyzed (Participants) | 15 | 9 | 22
  Month 12 | 0.1 (4.92) | 0.8 (1.64) | 0.7 (3.51)

11. Secondary Outcome: Absolute Value in Clinical Global Impression of Improvement (CGI-I) Score
Description: The Clinical Global Impression of Improvement (CGI-I) is a global measure of improvement or change based on the clinician's assessment of all available clinical data obtained from interviewing the participant. The CGI-I consists of a single 7-point rating of total improvement or change from baseline severity, regardless of whether or not the change is due entirely to drug treatment. Raters select 1 response based on the following question, "Compared to your participant's condition at the beginning of treatment, how much has he/she changed?" Scores are: 1: Very much improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; or 7: Very much worse.
Time Frame: Month 6 and Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
Number analyzed (Participants) | 50 | 70 | 62
units on a scale
  Month 6: number analyzed (Participants) | 33 | 39 | 41
  Month 6 | 3.9 (1.04) | 4.2 (1.03) | 3.7 (1.19)
  Month 12: number analyzed (Participants) | 15 | 9 | 22
  Month 12 | 3.5 (1.30) | 4.6 (1.13) | 4.0 (1.21)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 20 mg PF-02545920 | 5 mg PF-02545920 Titration up to 20 mg | Placebo and Titration up to 20 mg PF-02545920
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/71 | 0/66
Serious Adverse Events (participants affected / at risk) | 7/51 | 9/71 | 5/66
Other Adverse Events (participants affected / at risk) | 32/51 | 53/71 | 54/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg PF-02545920 (N=51) | 5 mg PF-02545920 Titration up to 20 mg (N=71) | Placebo and Titration up to 20 mg PF-02545920 (N=66)
Huntington's disease (Congenital, familial and genetic disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Complication associated with device (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chorea (Nervous system disorders) | 0 | 1 | 0
Hyperkinesia (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg PF-02545920 (N=51) | 5 mg PF-02545920 Titration up to 20 mg (N=71) | Placebo and Titration up to 20 mg PF-02545920 (N=66)
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 4
Nausea (Gastrointestinal disorders) | 2 | 9 | 8
Vomiting (Gastrointestinal disorders) | 1 | 5 | 3
Fatigue (General disorders) | 2 | 9 | 9
Viral upper respiratory tract infection (Infections and infestations) | 4 | 3 | 7
Fall (Injury, poisoning and procedural complications) | 6 | 15 | 8
Weight decreased (Investigations) | 3 | 7 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 2 | 4
Chorea (Nervous system disorders) | 11 | 11 | 14
Dizziness (Nervous system disorders) | 0 | 9 | 5
Dyskinesia (Nervous system disorders) | 1 | 3 | 6
Headache (Nervous system disorders) | 1 | 5 | 3
Hyperkinesia (Nervous system disorders) | 7 | 0 | 2
Sedation (Nervous system disorders) | 1 | 2 | 5
Somnolence (Nervous system disorders) | 1 | 4 | 9
Anxiety (Psychiatric disorders) | 2 | 5 | 7
Depression (Psychiatric disorders) | 3 | 3 | 5
Insomnia (Psychiatric disorders) | 2 | 4 | 9
Restlessness (Psychiatric disorders) | 1 | 2 | 5
Sleep disorder (Psychiatric disorders) | 3 | 3 | 2

LIMITATIONS AND CAVEATS:
This study was terminated on 15 December 2016 due to study A8241021 showing no significant difference on primary endpoint between PF-02545920 and placebo. No safety concerns were associated with this termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT02342548/SAP_000.pdf
  • Study Protocol (2014-10-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02342548/Prot_001.pdf